CLINICAL TRIAL: NCT02859870
Title: Evaluation of the Colonoscope With Vision to 330 ° (Full Spectrum Endoscopy) in the Detection of Colorectal Adenomas
Acronym: FUSETM-Colon
Status: Completed | Type: Observational
Sponsor: Institut Paoli-Calmettes (Other)
Responsible Party: Sponsor
Other Study IDs: FUSE-TM-Colon-IPC 2015-002
Record Dates: First submitted 2016-08-02; First posted 2016-08-09 (Estimated); Last update posted 2017-08-21 (Actual); Status verified 2017-08

CONDITIONS: Colorectal Adenoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: FUSE-TM colonoscope — Colonoscopy in conditions of normal security including patient clinical examination before leaving the hospital. Data collection by each operator.

SUMMARY:
The coloscopy is considered as the gold standard for screening and resection of colorectal adenomas. However the literature reports that the rate of omitted adenoma is still high (24 to 41%). The development of the FUSE system (Endochoice, USA) allows a larger field of view with a projection onto 3 screens (330° vision). A pilot study and a randomized multicentre has demonstrated the feasibility with a significant improvement of the rate of detected adenomas. This first study in France concerning this technology has the objectives to demonstrate the feasibility in France, the safety and to compare the rate of detected adenomas with data of the literature.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years
* Diagnostic colonoscopy

Exclusion Criteria:

* Colorectal cancer
* Colic surgery
* Preparation of average or poor quality
* Rectal polyp of hyperplastic type <2 mm

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient with colorectal adenoma candidate to colonoscopy of diagnostic
Sampling Method: Non-Probability Sample
Enrollment: 141 (Actual)
Dates: Start 2015-03-18 (Actual); Primary Completion 2016-04-30 (Actual); Study Completion 2016-04-30 (Actual)

PRIMARY OUTCOMES:
Efficacy | 1 day
  Cecal intubation rate
Efficacy | 1 day
  Absence of necessity to change of endoscope in case of progression, visualization, biopsy or resection

SECONDARY OUTCOMES:
Toxicity | 1 day
  Serious adverse events (perforation, uncontrolled bleeding)

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Philippe RATONE, MD, Study Director — Institut Paoli-Calmettes
Locations (1):
- Institut Paoli Cakmettes, Marseille, Bouches du Rhône, France

REFERENCES:
- [Background] Gralnek IM, Segol O, Suissa A, Siersema PD, Carr-Locke DL, Halpern Z, Santo E, Domanov S. A prospective cohort study evaluating a novel colonoscopy platform featuring full-spectrum endoscopy. Endoscopy. 2013 Sep;45(9):697-702. doi: 10.1055/s-0033-1344395. Epub 2013 Aug 12. PMID 23939509
- [Background] Gralnek IM, Siersema PD, Halpern Z, Segol O, Melhem A, Suissa A, Santo E, Sloyer A, Fenster J, Moons LM, Dik VK, D'Agostino RB Jr, Rex DK. Standard forward-viewing colonoscopy versus full-spectrum endoscopy: an international, multicentre, randomised, tandem colonoscopy trial. Lancet Oncol. 2014 Mar;15(3):353-60. doi: 10.1016/S1470-2045(14)70020-8. Epub 2014 Feb 20. PMID 24560453
- [Background] Rex DK, Cutler CS, Lemmel GT, Rahmani EY, Clark DW, Helper DJ, Lehman GA, Mark DG. Colonoscopic miss rates of adenomas determined by back-to-back colonoscopies. Gastroenterology. 1997 Jan;112(1):24-8. doi: 10.1016/s0016-5085(97)70214-2. PMID 8978338
- [Background] Rex DK, Rahmani EY, Haseman JH, Lemmel GT, Kaster S, Buckley JS. Relative sensitivity of colonoscopy and barium enema for detection of colorectal cancer in clinical practice. Gastroenterology. 1997 Jan;112(1):17-23. doi: 10.1016/s0016-5085(97)70213-0. PMID 8978337
- [Background] Siersema PD, Rastogi A, Leufkens AM, Akerman PA, Azzouzi K, Rothstein RI, Vleggaar FP, Repici A, Rando G, Okolo PI, Dewit O, Ignjatovic A, Odstrcil E, East J, Deprez PH, Saunders BP, Kalloo AN, Creel B, Singh V, Lennon AM, DeMarco DC. Retrograde-viewing device improves adenoma detection rate in colonoscopies for surveillance and diagnostic workup. World J Gastroenterol. 2012 Jul 14;18(26):3400-8. doi: 10.3748/wjg.v18.i26.3400. PMID 22807609